CLINICAL TRIAL: NCT06027229
Title: Additional Recombinant COVID-19 Humoral and Cell-Mediated Immunogenicity in Immunosuppressed Populations
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Novavax (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2023-1208; Protocol Version 10/5/2024 (Other: UW Madison); SMPH/MEDICINE/GASTROENT (Other: UW Madison); A534250 (Other: UW Madison)
Record Dates: First submitted 2023-08-31; First posted 2023-09-07 (Actual); Results first posted 2025-10-20 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-04

CONDITIONS: Immunosuppression; COVID-19
Keywords: Immunogenicity; IBD; solid organ transplant
MeSH Terms: conditions — COVID-19 | interventions — NVX-CoV2373 adjuvated lipid nanoparticle

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Participants who have had Solid Organ Transplants (Experimental): Male and females aged 18 to 85 who are solid organ transplant recipients and receive the study intervention.
  Interventions: Biological: NVX-CoV2372
- Participants with IBD (Experimental): Male and females aged 18 to 85 who have IBD and receive the study intervention.
  Interventions: Biological: NVX-CoV2372

INTERVENTIONS:
Biological: NVX-CoV2372 — Novavax COVID-19 Vaccine Booster for Omicron XBB.1.5
  Other Names: Novavax COVID-19 Vaccine

SUMMARY:
To determine whether providing a recombinant booster COVID-19 vaccine improves sustained humoral and cell-mediated immunogenicity against SARS-CoV-2 in immunosuppressed patients with Inflammatory Bowel Disease (IBD) and/or solid organ transplant recipients. 120 participants will be enrolled and can expect to be on study for 6 months.

DETAILED DESCRIPTION:
This will be a single-center, prospective, unblinded, non-randomized study of 120 immunosuppressed patients who are planning to receive a recombinant COVID-19 vaccine booster dose as standard of care and are willing to participate in the study. At least 35 patients will have inflammatory bowel disease and at least 35 patients will be a solid organ transplant recipient. After obtaining informed consent, individuals who meet the inclusion criteria and none of the exclusion criteria will be invited to participate in the study. Blood samples will be collected from each participant at the baseline visit (V1), at 1 month post-booster (V2 visit), and 6 months post-booster (V3).

Aim 1: To determine whether providing a recombinant booster COVID-19 vaccine improves sustained humoral and cell-mediated immunogenicity against SARS-CoV-2 in immunosuppressed patients with IBD and/or solid organ transplant recipients.

The investigators hypothesize that solid organ transplant recipients receiving a combination of immunosuppressive regimens will have lower antibody concentrations than patients with IBD because previous work has shown that patients with IBD have higher rates of seroconversion than solid organ transplant recipients.

Per Protocol Amendment Approved 10/23/24: The 2024-2025 season activities will not proceed as originally planned due to the withdrawal of financial support. Study will be completed with 21 participants per updated analyses.

ELIGIBILITY:
Inclusion Criteria:

• Patient has a history of ulcerative colitis (UC), Crohn's disease, pouchitis, or indeterminate colitis diagnosed by standard clinical, radiographic, endoscopic, and histopathologic criteria.

And / or patient is a solid organ transplant recipient (e.g. lung, kidney, liver)

* Have received at least three doses of a COVID-19 vaccine.

  * Three messenger RNA (mRNA) vaccines, or
  * One or two viral vector vaccine and one or two mRNA vaccines.
* Female participant of non-childbearing potential (pre-menarche, current tubal ligation, hysterectomy, oophorectomy or post-menopause) and childbearing potential (if they had: practiced adequate contraception for 1 month prior to vaccination and agreement to use such for an additional 8 weeks after administration of the Novavax COVID-19 vaccine). Non-pregnant females with a negative pregnancy test who are willing to practice adequate contraception 8 weeks after administration of the Novavax COVID-19 vaccine.
* On one of the following treatment regimens

  * IBD

    * Thiopurine Therapy Group: on azathioprine at least 2.0mg/kg or 6MP 1.0mg/kg
    * Anti-TNF Therapy Group: on maintenance therapy infliximab (at least 8 every 8 weeks), golimumab (at least monthly), adalimumab (at least every 2 weeks), or certolizumab (at least monthly)
    * Anti-TNF Combination Therapy Group: on anti-TNF therapy as described above along with either 15mg of methotrexate or azathioprine at least 1.0mg/kg or 6MP 0.5mg/kg.
    * Vedolizumab Therapy Group: either vedolizumab monotherapy at least every 8 week dosing or combination therapy Group: on vedolizumab therapy at with azathioprine or methotrexate
    * Ustekinumab Therapy Group: either ustekinumab monotherapy or combination therapy with methotrexate or azathioprine.
    * Tofacitinib Therapy Group: on tofacitinib at least 5mg orally, twice per day
    * Risankizumab Therapy: 360mg at least every 8 weeks
    * Upadactinib Therapy Group: on upadactinib at least 15mg orally
    * Ozanimod: 0.92mg once daily
  * Solid organ transplant recipient (on any dose of the following regimens: patients can be on more than one of the regimens below)

    * Mycophenolate
    * Tacrolimus or cyclosporine
    * Sirolimus or everolimus
    * Azathioprine
    * Corticosteroids
    * Belatacept

Exclusion Criteria:

* Allergy to recombinant COVID-19 vaccine or any component of it
* Patient cannot or will not provide written informed consent.
* Unable to provide appropriate informed consent because of illiteracy or impairment in decision-making capacity.
* Active antibody-mediated or cellular rejection within the past six months
* Recent IBD flare requiring initiation of systemic corticosteroids within the past month.
* Previous history of myocarditis or pericarditis ever.
* Patients who are pregnant
* Patients who are lactating
* Patients with an active COVID-19 infection
* Patients with a COVID-19 infection within the past two months

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2023-11-20 (Actual); Primary Completion 2024-04-24 (Actual); Study Completion 2024-09-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Freddy Caldera, DO, MS, Principal Investigator — UW School of Medicine and Public Health
Locations (1):
- UW School of Medicine and Public Health, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 21 participants were assessed for eligibility, 1 patient was withdrawn due to inadvertent administration of an messenger ribonucleic acid (mRNA) vaccine.
Groups:
- Immunosuppressed Participants: Male and females aged 18 to 85 who are solid organ transplant recipients or have Irritable Bowel Disease (IBD) and receive the study intervention.
  NVX-CoV2372: Novavax COVID-19 Vaccine Booster for Omicron XBB.1.5
Period: Overall Study
Arm/Group | Immunosuppressed Participants
Started | 20
Follow-Up | 20
Analysis Population | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Immunosuppressed Participants: Male and females aged 18 to 85 who are solid organ transplant recipients or have IBD and receive the study intervention.
  NVX-CoV2372: Novavax COVID-19 Vaccine Booster for Omicron XBB.1.5
Arm/Group | Immunosuppressed Participants
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.6 (14.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 20
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilograms per meter squared] | 79.59 (10.2)
Smoking Status [Count of Participants; unit: Participants]
  Never | 14
  Former | 6
  Current | 0
Type of Immunosuppression [Count of Participants; unit: Participants]
  IBD | 17
  Solid Organ Transplantation | 3
Type of IBD [Count of Participants; unit: Participants] — Population: Only participants with IBD are counted in this measure.
  Participants
    Proctitis: number analyzed (Participants) | 17
    Proctitis | 1
    Proctosigmoiditis: number analyzed (Participants) | 17
    Proctosigmoiditis | 1
    Left Sided Disease: number analyzed (Participants) | 17
    Left Sided Disease | 1
    Pancolitis: number analyzed (Participants) | 17
    Pancolitis | 2
Previous Surgical Resection [Count of Participants; unit: Participants] | 6
Length of IBD [Mean (Standard Deviation); unit: years] — Population: Only participants with IBD are counted in this measure.
  years
    number analyzed (Participants) | 17
    (all) | 16 (12.2)
Current IBD Medications [Count of Participants; unit: Participants] — Population: 17 participants have IBD
  Participants
    Azathioprine: number analyzed (Participants) | 17
    Azathioprine | 1
    Metho: number analyzed (Participants) | 17
    Metho | 2
    Remicade: number analyzed (Participants) | 17
    Remicade | 4
    Humira: number analyzed (Participants) | 17
    Humira | 4
    Entyvio: number analyzed (Participants) | 17
    Entyvio | 5
    Stelara: number analyzed (Participants) | 17
    Stelara | 2
    Xeljanz: number analyzed (Participants) | 17
    Xeljanz | 1
    Skyrizi: number analyzed (Participants) | 17
    Skyrizi | 1
Type of Transplant [Count of Participants; unit: Participants] — Population: 3 participants had solid organ transplant
  Participants
    Liver: number analyzed (Participants) | 3
    Liver | 1
    Lung: number analyzed (Participants) | 3
    Lung | 2
Current Transplantation Medications [Count of Participants; unit: Participants] — Population: 3 participants had solid organ transplant
  Participants
    Prednisone: number analyzed (Participants) | 3
    Prednisone | 2
    Azathioprine: number analyzed (Participants) | 3
    Azathioprine | 1
    Tacrolimus: number analyzed (Participants) | 3
    Tacrolimus | 3
    Mycophenolate: number analyzed (Participants) | 3
    Mycophenolate | 2
History of COVID-19 infection [Count of Participants; unit: Participants]
  Never | 9
  Once | 8
  Twice | 2
  Thrice | 1
Number of COVID-19 Vaccines Received [Mean (Full Range); unit: vaccinations] | 4.7 [3 to 8]

OUTCOME MEASURES:

1. Primary Outcome: Change in Antibody Concentration From Baseline (Visit 1) at 1 Month (Visit 2)
Description: Antibody concentrations 1 month after the recombinant vaccine booster (V2) in patients with IBD and solid organ transplant recipients compared to their baseline visit (V1).
Time Frame: baseline and 1 month
Measure: Mean (95% Confidence Interval); unit: Endotoxin Units per milliliter (EU/mL)
Arm/Group | Immunosuppressed Participants
Number analyzed (Participants) | 20
Endotoxin Units per milliliter (EU/mL)
  baseline | 22968.5 [12081.4 to 43666.4]
  1 month | 66639 [37915.5 to 117124.0]

2. Secondary Outcome: Seropositivity Rates
Description: Seropositive will be defined by positive anti-receptor binding domain (RBD) IgG antibodies specific to SARS-CoV-2 performed by Labcorp.
Time Frame: baseline, 1 month, 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Immunosuppressed Participants
Number analyzed (Participants) | 20
Participants
  baseline | 20
  1 month | 20
  6 months | 20

3. Secondary Outcome: Percent of Participants Seronegative at Baseline and Subsequently Seropositive
Description: Percentages (and 2-sided 95% Confidence Intervals) of participants who were seronegative at baseline and became seropositive after immunization will be evaluated in each group. For initially seropositive subjects at V1, antibody concentration at post-vaccination (V2) ≥ 4 fold the pre-vaccination antibody concentration.
Time Frame: baseline, 1 month, 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Immunosuppressed Participants
Number analyzed (Participants) | 20
Participants
  baseline | 0
  1 month | 0
  6 months | 0

4. Secondary Outcome: Change in Interferon Gamma Responses at 1 Month Compared to Baseline
Description: An interferon gamma response will be considered any measurable response, reported is change in cells per million from baseline to 1 month.
Time Frame: baseline and 1 month
Measure: Mean (Standard Deviation); unit: cells per million
Arm/Group | Immunosuppressed Participants
Number analyzed (Participants) | 20
cells per million | 28 (101)

5. Secondary Outcome: Change in Interferon Gamma Responses at 6 Months Compared to 1 Month
Description: An interferon gamma response will be considered any measurable response, reported is change in cells per million from 1 month to 6 months.
Time Frame: 1 month, 6 months
Measure: Mean (Standard Deviation); unit: cells per million
Arm/Group | Immunosuppressed Participants
Number analyzed (Participants) | 20
cells per million | -0.625 (164)

6. Secondary Outcome: Solicited Adverse Events (AEs)
Description: The number of participants reporting each solicited local AE and each solicited systemic AE within seven days (Days 1-7) after the booster dose and overall will be summarized.
  * Solicited local AEs included injection site pain, redness, and swelling.
  * Solicited systemic AEs included fatigue, myalgia, arthralgia, headache, shivering/chills, fever, and gastrointestinal symptoms (nausea, vomiting, diarrhea, and abdominal pain).
Time Frame: up to 7 days on study
Measure: Count of Participants; unit: Participants
Arm/Group | Immunosuppressed Participants
Number analyzed (Participants) | 20
Participants | 12

7. Secondary Outcome: Unsolicited Adverse Events
Description: The number of participants reporting unsolicited AEs within 30 days (Days 1-30) after the booster dose and overall will be summarized for both the study groups.
Time Frame: up to 30 days on study
Measure: Count of Participants; unit: Participants
Arm/Group | Immunosuppressed Participants
Number analyzed (Participants) | 20
Participants | 1

8. Secondary Outcome: Potential Immune-Mediated Diseases (pIMDs)
Description: The number of participants reporting pIMDs from the booster dose to the study end will be summarized.
Time Frame: up to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Immunosuppressed Participants
Number analyzed (Participants) | 20
Participants | 0

9. Secondary Outcome: Serious Adverse Events (SAEs)
Description: The number of participants reporting SAEs and fatal SAEs from the booster dose administration to the study end will be summarized for both the study groups.
Time Frame: up to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Immunosuppressed Participants
Number analyzed (Participants) | 20
Participants | 0

10. Secondary Outcome: Number of Participants Reporting Disease Flares of IBD
Description: Disease activity will be assessed by monitoring disease activity using the Short Crohn's Activity Index (SCAI)18 for patients with Crohn's disease or the Simple Clinical Colitis Activity Index (SCCAI) questionnaire for patients with Ulcerative colitis at the baseline visit (V1), V2, and V3 visits. The incidence of IBD flares will be evaluated in all patients receiving recombinant boosters. This will be quantified by patients who were in clinical remission who develop a disease flare after receiving a recombinant COVID-19 booster.
Time Frame: up to 6 months
Population: 17 participants had IBD
Measure: Count of Participants; unit: Participants
Arm/Group | Immunosuppressed Participants
Number analyzed (Participants) | 17
Participants | 0

11. Secondary Outcome: Number of Participants Reporting Acute Rejection of Their Transplant
Description: Participants will be asked if they have been diagnosed with acute rejection after their baseline visit (V1). Episodes of acute rejection will be collected by searching electronic medical records and asking patients at each clinic visit (V2 and V3). Acute rejection will be defined as a notation of a new episode of acute rejection (cellular or antibody-mediated), a steroid bolus and taper in the absence of another indication, or administration of a T or B cell depleting agent or immune globulin. This will be quantified by patients who were who developing acute rejection of their transplant after receiving a recombinant COVID-19 booster.
Time Frame: up to 6 months
Population: 3 participants had solid organ transplants
Measure: Count of Participants; unit: Participants
Arm/Group | Immunosuppressed Participants
Number analyzed (Participants) | 3
Participants | 0

ADVERSE EVENTS:
Time Frame: up to 180 days post-booster
Description: Participants were instructed to contact the study team if they experienced fever, chills, or rash. 7 days after each vaccination, participants were contacted to assess for solicited adverse events and to document any unsolicited adverse events. Local reactions (e.g., injection site pain, redness, swelling) and systemic symptoms (e.g., fever, headache, fatigue, myalgia) were recorded for 7 days following each dose, while unsolicited adverse events were monitored for 30 days.
Arm/Group | Immunosuppressed Participants
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 12/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Immunosuppressed Participants (N=20)
Injection Site Pain (Injury, poisoning and procedural complications) | 8
Headache (General disorders) | 10
Paresthesia (General disorders) | 1
Gastrointestinal Symptoms (General disorders) | 4
Shivering or Chills (General disorders) | 2
Arthralgia (General disorders) | 9
Myalgia (General disorders) | 5
Fatigue (General disorders) | 8
Injection Site Swelling (Injury, poisoning and procedural complications) | 1
Hematemesis (Gastrointestinal disorders) | 1
Hematochezia (Gastrointestinal disorders) | 1
Hematuria (Renal and urinary disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-10-05): https://cdn.clinicaltrials.gov/large-docs/29/NCT06027229/Prot_SAP_000.pdf